CLINICAL TRIAL: NCT00231205
Title: TDI-Derived Myocardial Preejection Velocities in Patients With Chronic Ischemic Left Ventricular Dysfunction Undergoing Surgical Revascularization
Brief Title: TDI Preejection Velocities and Myocardial Viability
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government); Czech Ministry of Education (Other Government)
Other Study IDs: IGA 8524-5
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2005-10-04 (Estimated); Status verified 2005-09

CONDITIONS: Coronary Artery Disease
Keywords: viability; myocardium; preejection velocity; CAD; echocardiography; tissue Doppler
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Revascularization

SUMMARY:
The purpose of the study is to test accuracy of positive preejection velocity to predict left ventricular remodeling and long-term prognosis after revascularization in 200 patients with chronically dysfunctional myocardium. Patients will be followed for 3 years.

Our hypothesis is that tissue-Doppler-derived analysis of positive preejection velocity allows to select optimal responders to revascularization; it means individuals with the greatest benefit in terms of LV remodeling and long-term prognosis.

DETAILED DESCRIPTION:
The objective of the project is to study clinical and prognostic value of new echocardiographic technique, so called positive preejection velocity (+VIC), in patients with chronic ischemic left ventricular (LV) dysfunction indicated for revascularization. Pilot studies has shown high accuracy of pulsed Tissue Doppler imaging (TDI)-derived resting pattern of +VIC to detect viable myocardium in patients with both acute myocardial infarction and chronically dysfunctional myocardium. The aim of the project is to test accuracy of +VIC to predict LV remodeling and long-term prognosis after revascularization in patients with chronically dysfunctional myocardium. Study population will consist of two groups of patients with stable ischemic LV dysfunction: group A- patients indicated for revascularization (n=200), group B- matched control group treated conservatively (case-control design) (n=100). All patients will be followed for 3 years. Endpoints include: 1) LV remodeling at 6 and 24 months and 2) MACE at 6, 12 and 36 months follow-up. Our hypothesis is that TDI-derived analysis of +VIC allows to select optimal responders to revascularization; it means individuals with the greatest benefit in terms of LV remodeling and long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. occluded or suboccluded left anterior descending coronary artery (LAD) at recent coronary angiography (< 3 months);
2. LV ejection fraction < 40%;
3. 3 and more akinetic or severely hypokinetic segments in the LAD perfusion territory at resting echocardiography.

Exclusion Criteria:

- Patients with recent acute coronary syndrome, atrial fibrillation, bundle branch block, LV hypertrophy or aneurysm, significant valvular disease, pacemakers or internal defibrillators, poor echocardiographic image quality and contraindications for MRI are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-01; Study Completion 2009-12

CONTACTS AND LOCATIONS:
Overall Officials: Martin Penicka, MD, PhD, Principal Investigator — Charles University, Prague, Czech Republic
Locations (1):
- III. Internal-cardiological clinic, 3rd Medical Faculty, Charles University, Prague, Czechia